CLINICAL TRIAL: NCT01647373
Title: Axial Length Change in Eyes Treated by Silicone Sponge Scleral Buckling.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0125-12
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2013-06-12 (Estimated); Status verified 2012-07

CONDITIONS: Rhegmatogenous Retinal Detachment
Keywords: retinal detachment; scleral buckle; silicone sponge; axial length; surgery included silicone sponge scleral buckling; retina currently attached; at least 6 months after surgery
MeSH Terms: conditions — Retinal Detachment

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
All existing medical literatue regarding axial length (AL) changes after scleral buckling surgery for retinal detachment, descibes changes after solid silicone buckling. In this hospital, the investigators use only silicone sponge buckling, which has different properties and a different buckle profile. there are no studies in the literature describing tha AL changes after sponge buckling, or whether the AL change is less or more than with solid silicone buckles. The investigators wish to determine whether the AL change profile with their silicone sponge is significantly different, and if so, whether this is clinically important in determining the better choice of buckle material to be preferred.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 6 months after succesful retinal detachment surgery
* with silicone sponge scleral buckling
* currently attached
* with IOL Master pre-surgery Axial Length measurement

Exclusion Criteria:

* patients with failed surgery and currently detached
* patients with vitreos silicone oil tamponade
* patients with radial or other non-circumference buckles
* patients with unclear media not amenable to IOL Master exam

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at least 6 months after succesful retinal detachment surgery, with silicone sponge scleral buckling, currently attached, and with IOL Master pre-surgery Axial Length measurement .
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-07 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Axial length in eye as measured by Zeiss IOL Master. | Single non-invasive measurement at 1 time point.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Rubowitz, MD, Principal Investigator — Retina Service, Meir Hospital
Locations (2):
- Israel (2):
  - Meir hospital, dept. Of ophthalmology, Kfar Saba
  - Retina Service, Meir Hospital, Kfar Saba